CLINICAL TRIAL: NCT00718497
Title: Comparing The Cyberlink Control System to the Manual Letter Board for Communication Purposes in the ALS Patient Population
Status: Completed | Type: Observational
Sponsor: Drexel University College of Medicine (Other)
Collaborators: MDA/ALS Center of Hope (Other)
Responsible Party: Sponsor
Organization: Drexel University (Other)
Other Study IDs: Internal-17018
Record Dates: First submitted 2008-07-14; First posted 2008-07-18 (Estimated); Last update posted 2013-03-05 (Estimated); Status verified 2013-03

CONDITIONS: Amyotrophic Lateral Sclerosis; Neurodegenerative Disease; Motor Neuron Disease
Keywords: Amyotrophic Lateral Sclerosis; Cerebrospinal Fluid; Neurodegenerative Disease; Motor Neuron Disease; Autonomic Nervous System; Neurodegenerative Diseases; Movement Disorders
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Neurodegenerative Diseases; Motor Neuron Disease; Movement Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- ALS: Subjects having either definite or probable ALS by El Escorial Criteria.

SUMMARY:
New technologies are giving people with motor disabilities alternative communication and control channels. The investigators are interested in using the Cyberlink Control System as a hands free means to access a computer for people with Amyotrophic Lateral Sclerosis (ALS). The goal of this project is to determine whether this device is a practical and realistic means for ALS patients to communicate with only the use of facial muscle, brainwave, and eye movements.

The benefit of this study may be of substantial value to many people with severe motor impairment. Additionally, it is hoped that some of the study subjects may benefit by incorporating hands-free computer use into their daily lives.

This study is intended to evaluate the effectiveness of the cyberlink as a tool for daily communication compared to the standard manual letter board.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of definite or possible ALS by the El Escorial Criteria
* Between ages of 18 to 89 years.
* Scored two or less in the ALS FRS category 1 (Speech)
* Scored two or less in the ALS FRS category 4 (Handwriting)
* Cognitively intact with no other neurological diseases
* No unstable medical problems

Exclusion Criteria:

* Any subject not meeting the inclusion criteria
* Patients unable to give informed consent either themselves or via a legally authorized personnel.
* Patients diagnosed with neurological problems other than ALS (upon examination by the principal investigator)

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ALS clinic patients at MDA/ALS Center of Hope.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2007-08; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Time Taken to Complete a Sentence | 1 session

CONTACTS AND LOCATIONS:
Overall Officials: Terry Heiman-Patterson, MD, Principal Investigator — MDA/ALS Center of Hope
Locations (1):
- MDA/ALS Center of Hope, Philadelphia, Pennsylvania, United States